CLINICAL TRIAL: NCT04677270
Title: Evaluation of Two Versions of a Digital Problem Solving Tool for the General Public Specific for the COVID-19 Pandemic
Acronym: COVIDPROBLEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Martin Kraepelien, Licensed clinical psychologist, Principal investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COVIDPROBLEM
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Problem Solving

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional interface (Experimental): Digital problem solving tool with a simple textbased graphical interface
  Interventions: Behavioral: Digital problem solving tool
- Advanced interface (Experimental): Digital problem solving tool with an advanced graphical interface and automatic functions
  Interventions: Behavioral: Digital problem solving tool

INTERVENTIONS:
Behavioral: Digital problem solving tool — Digital problem solving tool - adapted for practical and emotional problems during the COVID-19 pandemic

SUMMARY:
A digital problem solving tool was tailored to people in the general public with practical or emotional problems during COVID-19. Content analysis were used to account for the types of problems participants used the tool to solve. Participants were randomized to one of two versions of the problem solving tool, a simple and a more advanced graphical interface. These versions were compared on participant-rated usability, credibility and the level of actual interaction with the tool.

ELIGIBILITY:
Inclusion Criteria:

* can use the Swedish language
* access to, and knowledge how to use, a digital internet-capable device

Exclusion Criteria:

* under 16 years
* no practical or emotional problems during pandemic

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | immediately after the intervention
  Self-rated assessment of usability, higher score is better
Treatment Credibility Scale | immediately after the intervention
  Self-rated assessment of treatment credibility, higher score is better

SECONDARY OUTCOMES:
Use of intervention | immediately after the intervention
  How much has the participant interacted with the problem solving tool.

OTHER OUTCOMES:
Problem categories | immediately after the intervention
  What categories of problems do participants solve with the problem solving tool.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kraepelien, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Centrum för Psykiatriforskning, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hentati A, Forsell E, Ljotsson B, Kraepelien M. Practical and Emotional Problems Reported by Users of a Self-guided Digital Problem-solving Intervention During the COVID-19 Pandemic: Content Analysis. JMIR Form Res. 2021 Oct 4;5(10):e31722. doi: 10.2196/31722. PMID 34559670